CLINICAL TRIAL: NCT02830360
Title: Ventricular Tachycardia Antiarrhythmics or AblatioN In Structural Heart Disease 2
Brief Title: Antiarrhythmics or Ablation for Ventricular Tachycardia 2
Acronym: VANISH2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John Sapp (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Abbott Medical Devices (Industry); Biosense Webster, Inc. (Industry); Ottawa Heart Institute Research Corporation (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Cardiac Arrhythmia Network of Canada (Other); Abbott (Industry); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, John Sapp, Staff Physician, Division of Cardiology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAPP004
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: Antiarrhythmic drug therapy; VT Catheter ablation; ICD Therapy; Ischemic Heart Disease
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia | interventions — Amiodarone; Sotalol; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VT catheter ablation (Active Comparator): Catheter ablation of ventricular tachycardia
  Interventions: Procedure: Catheter ablation
- Antiarrhythmic Drug Therapy (Active Comparator): Patients will be prescribed either oral amiodarone or sotalol daily (dosage and frequency to be determined based on patient's clinical presentation at the time of the qualifying arrhythmia).
  Interventions: Drug: Antiarrythmic Drug Therapy

INTERVENTIONS:
Drug: Antiarrythmic Drug Therapy — Patients will be prescribed antiarrhythmic drugs (either amiodarone or sotalol based on specific clinical presentation, including medical history, functional class, ejection fraction, and renal function.)
  Other Names: Amiodarone (Cordarone) or Sotalol (Sotacor)
  Arms: Antiarrhythmic Drug Therapy
Procedure: Catheter ablation — Intracardiac electrode catheters are placed via central vasculature to identify myocardial scar, and surviving conduction channels within the scar which form the substrate for ventricular tachycardia. Radiofrequency energy is applied to these sites, interrupting the VT circuits.
  Other Names: VT ablation
  Arms: VT catheter ablation

SUMMARY:
A multicenter, randomized clinical trial to assess whether catheter ablation or antiarrhythmic drug therapy provides the most effective control of important clinical outcomes for patients with prior myocardial infarction and sustained monomorphic ventricular tachycardia (VT).

DETAILED DESCRIPTION:
Implantable Defibrillators (ICDs) reduce sudden death and can terminate some VT without shocks, but they don't prevent VT; the most appropriate strategy to suppress VT remains unknown. Two randomized clinical trials have suggested that catheter ablation can significantly reduce the incidence of subsequent VT in patients after an initial episode. Neither trial, however, compared catheter ablation to active antiarrhythmic drug therapy. Randomized trials of antiarrhythmic drug therapy have demonstrated that therapy with either sotalol or amiodarone can reduce recurrent VT. Both antiarrhythmic drug and ablation therapy suffer from imperfect efficacy and the potential for significant side-effects. No study has compared ablation to drug therapy for first-line treatment. The VANISH study which compared ablation to aggressive antiarrhythmic drug therapy for patients who have failed initial drug therapy was published in May 2016, and demonstrated that for patients with drug-refractory VT, catheter ablation was superior to escalation of antiarrhythmic drug therapy. Benefits were seen in the group which had VT despite amiodarone. Event rates were similar between amiodarone and sotalol for patients with VT occurring despite sotalol, who were randomized to either new initiation of amiodarone or catheter ablation. These results do not address the clinical question of the most appropriate first line therapy for suppression of VT in persons with prior myocardial infarction, an ICD and VT.

The trial hypothesis is: catheter ablation will, in comparison to antiarrhythmic drug therapy reduce the composite outcome of death at any time, appropriate ICD shock after 14 days, ventricular tachycardia storm after 14 days or treated sustained ventricular tachycardia below the detection rate of the ICD for patients with prior myocardial infarction and sustained monomorphic ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Prior Myocardial Infarction and
* One of the following VT events while not being treated with amiodarone, sotalol, or another class I or class III antiarrhythmic drug) within the last 6 months:

  * Sustained monomorphic VT documented on 12-lead ECG or rhythm strip terminated by pharmacologic means or DC cardioversion
  * ≥3 episodes of VT treated with antitachycardia pacing (ATP), at least one of which was symptomatic
  * ≥ 5 episodes of VT treated with antitachycardia pacing (ATP) regardless of symptoms
  * ≥1 appropriate ICD shocks,
  * ≥3 VT episodes within 24 hours

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Active ischemia (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of VT (e.g. drug-induced arrhythmia), had recent acute coronary syndrome within 30 days, coronary revascularization (<90 days bypass surgery, <30 days percutaneous coronary intervention), or have CCS functional class IV angina. Note that biomarker level elevation alone after ventricular arrhythmias does not denote acute coronary syndrome or active ischemia.
* Are ineligible to take the antiarrhythmic drug to which they would be assigned due to allergy, intolerance or contraindication
* Are known to have protruding left ventricular thrombus or mechanical aortic and mitral valves
* Have had a prior catheter ablation procedure for VT
* Presenting arrhythmia: polymorphic VT or ventricular fibrillation (VF)
* Are in renal failure (Creatinine clearance <15 mL/min), have NYHA Functional class IV heart failure, or a systemic illness likely to limit survival to <1 year
* Have had recent ST elevation myocardial infarction or non-ST elevation MI (< 30 days); note that biomarker elevation alone after ventricular arrhythmias does not denote MI.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 8 years (including pilot study data)
  Time to any death occurring at any time post randomization
Appropriate ICD shock at least 14 days post randomization | 8 years (including pilot study data)
  Time to first appropriate ICD shock after 14 days post randomization
VT storm at least 14 days post randomization | 8 years (including pilot study data)
  Time to 3 or more episodes of VT within 24 hours
Sustained VT requiring treatment at least 14 days post randomziation | 8 years (including pilot study data)
  Time to any sustained VT greater below the detection rate of the ICD requiring cardioversion (electrical or chemical) or manual ICD therapy at least 14 days post randomization

SECONDARY OUTCOMES:
All-cause mortality at any time | 8 years (including pilot study data)
  Time to any death occurring at any time post randomization
Appropriate ICD ATP at any time or after 14 days | 8 years (including pilot study data)
  any appropriate therapy delivered from the ICD at least 14 days post randomization
Appropriate shocks at any time or after 14 days | 8 years (including pilot study data)
  appropriate ICD shocks at any time post randomization
VT storm at any time or after 14 days | 8 years (including pilot study data)
  3 or more episodes of VT occurring within 24 hours at any time post randomization; including incessant VT
Sustained VT not treated by ICD at any time or after 14 days | 8 years (including pilot study data)
  any sustained VT greater than 30 seconds captured on a rhythm strip, monitor zone, holter monitor, or 12 lead ECG
Time to sustained VT treated with appropriate any type of manual cardioversion after 14 days | 8 years (including pilot study data)
  Any sustained VT greater than 30 seconds requiring manual cardioversion (ICD, external or pharmacologic)
Inappropriate ICD shocks at any time or after 14 days | 8 years (including pilot study data)
  all inappropriate shocks from the ICD at any time post randomization
Any ICD shock at any time or after 14 days | 6 years (including pilot study data)
  Both appropriate and inappropriate shocks from the ICD at any time post randomization
Any ventricular arrhythmia event at any time or after 14 days (composite of appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion) | 8 years (including pilot study data)
  All ventricular arrhythmias including a composite of: appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion), VT storm/incessant VT.
Number of ICD shocks (all cause) | 8 years (including pilot study data)
  the number of all shocks from any cause will be calculated
Number of Anti-tachycardia pacing (ATP) | 8 years (including pilot study data)
  The total of all ATP delivered from the ICD will be calculated
Number of ICD appropriate therapy | 8 years (including pilot study data)
  Total number of therapies which received appropriate ICD therapy
Number of VT storm events | 8 years (including pilot study data)
  Total number of VT storms (3 episodes of VT within 24 hours)/ incessant VT will be calculated
Number of sustained VT events | 8 years (including pilot study data)
  Total number of sustained VT (greater than 30 seconds)
Number of ventricular arrhythmia events | 8 years (including pilot study data)
  This is a composite of appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion, or VT storm/incessant VT. VT events which do not terminate despite exhausting ICD therapies will be considered incessant VT and included within the definition of VT storm.
Hospital admission for cardiac causes | 8 years (including pilot study data)
  Hospitalizations greater than 24 hours due to a cardiovascular cause.
Ablation procedural complications or antiarrhythmic drug adverse effects (this may require a separate substudy, depending on data complexity) | 8 years (including pilot study data)
  Periprocedural complications and adverse drug reactions will be assessed
Serious adverse events | 8 years (including pilot study data)
  Serious events is any event which causes death, hospitalization, is life threatening and is directly related to the study treatment.
Side effects from anti-arrhythmic medication | 8 years (including pilot study data)
  Any dose change or discontinuation of anti-arrhythmic medication due to abnormal blood tests (including kidney function, liver function, thyroid function) or any perceived side effects.
Quality of life - SF36 | 8 years (including pilot study data)
  Will include responses from the Short Form 36
Quality of life - EQ5D | 8 years (including pilot study data))
  Will include responses from the Euroquol 5D questionnaire
Quality of life - HADS | 8 years (including pilot study data)
  Will include responses from the Hospital Anxiety and Depression Scale quesionnaire
Cost-effectiveness | 8 years (including pilot study data)
  Quality adjusted life years (QALYs) will be derived from the case report forms and the questionnaires
Escalation and De-escalation of antiarrhythmic medication | 8 years (including pilot study data)
  Any increase or decrease in the dosage of antiarrhythmic medication either due to inefficacy or side effects will be assessed.
ICD Revision | 8 years (including pilot study data)
  Surgical revisions to implanted defibrillators at any time

CONTACTS AND LOCATIONS:
Overall Officials: John L Sapp, MD FRCPC, Principal Investigator — Nova Scotia Health Authority; Ratika Parkash, MD MSc FRCPC, Study Director — Nova Scotia Health Authoriry; Anthony L Tang, MD FRCPC, Study Director — London Health Sciences Centre; George A Wells, BSc MSc PhD, Study Director — Ottawa Heart Institute Research Corporation; William G Stevenson, MD, Study Director — Brigham and Women's Hospital; Jeff Healey, MD FRCPC, Study Director — Population Health Research Institute, McMaster University
Locations (22):
- United States (2):
  - Hartford General Hospital, Hartford, Connecticut
  - Vanderbilt University Hospital, Nashville, Tennessee
- Canada (18):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Interior Health Authority, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - Queen's University Health Sciences Centre, Kingston, Ontario
  - St. Mary's Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Universitaire de Montreal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - Institut Universitaire de cardiologie et pneumologie de Quebec - Laval University Hosptial, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- France (2):
  - Hopitaux de Bordeaux, Bordeaux, Acquitaine
  - CHU - University Hospital Nancy, Nancy, Meurthe-et-Moselle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nery PB, Wells GA, Tang ASL, Parkash R, Stevenson W, Healey JS, Gula L, Nair GM, Essebag V, Rivard L, Deyell MW, Sarrazin JF, Amit G, Roux JF, AbdelWahab A, Lane C, Samuel M, Sandila N, Sapp JL; VANISH2 Study Team. Catheter Ablation vs Sotalol or Amiodarone for Ventricular Tachycardia: A Substudy of the VANISH2 Trial. J Am Coll Cardiol. 2026 Jan 20;87(2):157-168. doi: 10.1016/j.jacc.2025.09.1595. Epub 2025 Oct 11. PMID 41217320
- [Derived] Sapp JL, Tang ASL, Parkash R, Stevenson WG, Healey JS, Gula LJ, Nair GM, Essebag V, Rivard L, Roux JF, Nery PB, Sarrazin JF, Amit G, Raymond JM, Deyell M, Lane C, Sacher F, de Chillou C, Kuriachan V, AbdelWahab A, Nault I, Dyrda K, Wilton S, Jolly U, Kanagasundram A, Wells GA; VANISH2 Study Team. Catheter Ablation or Antiarrhythmic Drugs for Ventricular Tachycardia. N Engl J Med. 2025 Feb 20;392(8):737-747. doi: 10.1056/NEJMoa2409501. Epub 2024 Nov 16. PMID 39555820
- [Derived] Sapp JL, Tang ASL, Parkash R, Stevenson WG, Healey JS, Wells G. A randomized clinical trial of catheter ablation and antiarrhythmic drug therapy for suppression of ventricular tachycardia in ischemic cardiomyopathy: The VANISH2 trial. Am Heart J. 2024 Aug;274:1-10. doi: 10.1016/j.ahj.2024.04.009. Epub 2024 Apr 21. PMID 38649085
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933